CLINICAL TRIAL: NCT03788486
Title: A Phase 4 Study to Assess the Clinical Efficacy and Safety of Meibomian Gland Dysfunction and Dry Eye With an LED Blue Light Treatment Device
Brief Title: Efficacy and Safety of Meibomian Gland Dysfunction and Dry Eye With an LED Blue Treatment Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid
Sponsor: Toyos Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCQ2019
Record Dates: First submitted 2018-12-25; First posted 2018-12-27 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Meibomian Gland Dysfunction
Keywords: dry eye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Single site prospective study with no control group to assess the safety and clinical efficacy of a low power LED light device on the signs and symptoms of dry eye disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2-3 Joule light device for MGD/Dry eye (Experimental): patients who qualify for the study will receive interventional in office treatments with the light treatment device in the upper and lower lids for defined periods of time twice weekly for a total of one month. Non-invasive tear break up, subjective questionnaires and corneal fluorescein staining will be measured through the course of the study.
  Interventions: Device: 2-3 Joule LED blue light device

INTERVENTIONS:
Device: 2-3 Joule LED blue light device — application of blue light LED light device for 2 minutes in the central lower lids, temporal lower lids and upper temporal lids twice weekly under observation for one month

SUMMARY:
This study will test the efficacy and safety of application of LED light to meibomian glands in upper and lower eyelids in eyes of patients suffering with meibomian gland disease.

DETAILED DESCRIPTION:
This study will test the efficacy and safety of application of LED light to meibomian glands in upper and lower eyelids in eyes of patients suffering with meibomian gland disease.

The primary objective of the study is to investigate the safety and efficacy of blue LED light with meibomian gland expression of the upper and lower eyelids in dry eye disease by change from baseline in subjective questionnaire and by measurement of non-invasive tear break up time.

Primary Endpoint: Improvement of tear break up time over the length of the study

Secondary endpoint: subjective patient comfort over the length of the study using a validated dry eye comfort questionnaire administered at each study visit, VAS, 0= no pain and 100 = maximal discomfort, Improvement in the number of corneal SPK that stain with fluorescein.

20 study subjects 18-85 will be enrolled with male or female in the Nashville and Memphis, TN areas who are generally healthy but have signs and symptoms of dry eye disease with Meibomian gland dysfunction.

phase 4

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form and HIPPA authorization.
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 -85.
4. Diagnosed with mild to severe dry eye in one or both eyes with evidence of Meibomian gland dysfunction: cloudy or thick secretions, lack of secretions or presence of telengiectasias on the lower lid margin.
5. History of persistent symptoms despite use of artificial tears.
6. Tear break up time of 7 seconds or less
7. Have normal lid anatomy.
8. Subject is able and willing to comply with the treatment, follow up schedule and requirements.
9. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 4 weeks after the end of the study.
10. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner
11. Are postmenopausal (no menstrual cycle for at least one year prior to Visit 1) or have undergone bilateral tubal ligation, hysterectomy, hysterectomy with uni- or bilateral oophorectomy, or bilateral oophorectomy.

    -

Exclusion Criteria:

1. Have a known hypersensitivity or contraindication to the investigational product or components.
2. Pregnancy or lactation
3. Subjects can be on the following medications if they have been on a stable dose for 12 weeks: topical cyclosporine, topical liftigrast and/or topical loteprednol etabonate. Tetracycline compounds, omega 3s, anticholinergics, anticonvulsants, antidepressants, retinoids, systemic immunosuppressive agents including oral corticosteroids, non-steroidals, antihistamines, or mast cell stabilizers, punctal plugs, contact lens wear and glaucoma medications.
4. Subjects must be unwilling to abstain from eyelash growth medications for the duration of the trial.
5. Subjects must not have had penetrating intraocular surgery, refractive surgery or corneal transplantation, eyelid surgery within 12 weeks prior to Visit 1.
6. Febrile illness within one week.
7. Treatment with another investigational drug or other intervention within one month.
8. Subjects with a history of herpetic keratitis.
9. Have serious or severe disease or uncontrolled medical condition that in the judgement of the investigator could confound study assessments or limit compliance.
10. Neuro-paralysis or pre-cancerous lesions in the area to be treated.
11. Radiation to the head or neck within past 12 months.
12. Planned radiation therapy or chemotherapy.
13. Anticipated relocation or extensive travel outside of the local study area preventing compliance with study procedures.
14. Legally blind in either eye.
15. Facial IPL treatment within 3 months of treatment.
16. Expression of Meibomian glands within 3 months prior to treatment.

    -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Estimated)

PRIMARY OUTCOMES:
change of non invasive tear break up time over the course of the study | one month
  3 measurements of non invasive tear break up time by investigator with average recorded

SECONDARY OUTCOMES:
subjective patient comfort as measured by validated VAS (visual analog scale) dry eye comfort questionnaire | one month
  patient completed questionnaire 10 mm in length minimum score 0=no pain and maximal score 100= maximal pain
change of number of corneal spk stained with fluorescein over the course of the study | one month
  manual counting of number of corneal spk

CONTACTS AND LOCATIONS:
Overall Officials: Rolando Toyos, MD, Study Chair — owner
Locations (2):
- United States (2):
  - Toyos Clinic, Germantown, Tennessee
  - Toyos Clinic, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
non-identifying patient data available upon request
Supporting Information: Study Protocol, ICF
Time Frame: one year beginning 6 months after study completion
Access Criteria: scientific researcher